CLINICAL TRIAL: NCT06816719
Title: A Randomized, Open-label, Single Dose, 2x4 Crossover Study to Evaluate the Safety and Pharmacokinetic Characteristics After Co-administration of JW0106 and C2101 and Administration of JW0107 in Healthy Volunteers Under Fasting Conditions
Brief Title: To Evaluate the Safety and PK Characteristics in Healthy Volunteers-JW24107
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: JW24107
Record Dates: First submitted 2025-01-01; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): (Period 1/3: Treatment A) (Period 2/4: Treatment B)
  Treatment A: JW0106 1 tablet + C2101 1 tablet Treatment B: JW0107 1 tablet
  Interventions: Drug: Treatment A: JW0106 1 tablet + C2101 1 tablet; Drug: Treatment B: JW0107 1 tablet
- Sequence 2 (Other): (Period 1/3: Treatment B) (Period 2/4: Treatment A)
  Treatment A: JW0106 1 tablet + C2101 1 tablet Treatment B: JW0107 1 tablet
  Interventions: Drug: Treatment A: JW0106 1 tablet + C2101 1 tablet; Drug: Treatment B: JW0107 1 tablet

INTERVENTIONS:
Drug: Treatment A: JW0106 1 tablet + C2101 1 tablet — * Co-administration of 1 tablet of JW0106 and 1 tablet of C2101
  * Administration orally with 150 mL of water under fasting conditions
Drug: Treatment B: JW0107 1 tablet — * Administration alone of 1 tablet of JW0107
  * Administration orally with 150 mL of water under fasting conditions
  Other Names: Administration alone of 1 tablet of JW0107

SUMMARY:
The objective is to evaluate the safety and pharmacokinetic characteristics after co-administration of JW0106 and C2101 and administration of JW0107 in healthy volunteers under fasting conditions.

DETAILED DESCRIPTION:
Pharmacokinetic characteristics: Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

Safety: All adverse events are summarized in terms of the number of subjects, expression rate, and number of expressions of adverse reactions by treatment group.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

Exclusion Criteria:

Subjects does not meet the inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
AUCt | Day 1(0 hour~12 hour), Day 2(24 hour), Day 3(48 hour), Day 4(72 hour)
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.
Cmax | Day 1(0 hour~12 hour), Day 2(24 hour), Day 3(48 hour), Day 4(72 hour)
  Describes the blood concentration statistically by pharmacokinetic blood

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Jeonbuk National University Hospital, Jeonju, Korea, South Korea